CLINICAL TRIAL: NCT03829189
Title: Interventional Study Comparing the Effect of a High-fiber Supplement Versus Placebo on the Body and the Brain
Brief Title: High-fiber Diet on the Body and the Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Max Planck Institute for Human Cognitive and Brain Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: GUT_BRAIN
Record Dates: First submitted 2019-01-11; First posted 2019-02-04 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Diet Modification; Overweight
Keywords: microbiome; food wanting; memory; fiber
MeSH Terms: conditions — Overweight | interventions — Inulin; maltodextrin

STUDY DESIGN:
Intervention Model Description: Arm 1: inulin; minimum of 14 days wash-out; 14 days placebo Arm 2: 14 days placebo; minimum of 14 days wash-out; 14 days placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inulin (Active Comparator)
  Interventions: Dietary Supplement: inulin
- maltodextrin (Placebo Comparator)
  Interventions: Dietary Supplement: maltodextrin

INTERVENTIONS:
Dietary Supplement: inulin — prebiotic supplement
  Arms: inulin
Dietary Supplement: maltodextrin — placebo supplement
  Arms: maltodextrin

SUMMARY:
The central research question aims to understand what drives individuals to make and maintain a vegan / vegetarian dietary decision, to investigate whether there are possible predictors that might influence such a decision and whether personality differences already exist or can only be measured after the change in diet. The investigators will examine the effects of a high-fiber diet on food wanting on a neural and on a behavioral level. The microbiome is suggested to mediate the expected changes in food wanting.

ELIGIBILITY:
Inclusion Criteria:

* body-mass-index 25-30kg/m^2
* females on contraception only

Exclusion Criteria:

* current neurological or psychiatric illness
* daily consumption of more than 50 g of alcohol, more than 10 cigarettes or more than 6 cups of coffee
* use of antidepressants or other centrally acting drugs
* type 2 diabetes mellitus or other serious metabolic disorders
* MRI contraindication (e.g. cardiac pacemaker, drug pump, shunts)
* major untreated medical condition, including gastrointestinal organs, lungs, heart, cardiovascular system, liver and kidney)
* diet-related restrictions (food allergies, food intolerances, known nutrient deficiencies or a recent history of dieting or restrictive eating behaviour, including vegan, vegetarian diet)
* current pregnancy or lactation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
fMRI BOLD activity during food wanting | 14 days
microbial alpha and beta diversity | 14 days
  The taxonomic structure of the microbial community will be determined using 16S rRNA gene sequencing. The reads from the sequencing data will be assigned to taxa by sequence similarity using puplic available data bases. Relative distribution of microbial taxa is then based on the number of reads assigned to each taxa. For the description of the the community the alpha diversity of each sample will be determined based on species richness, evenness of species distribution which is combined in the single value of the Shannon diversity index. Furthermore beta-diversity, how the microbial communities differ between sample, will be analysed by principal component analysis as well as non-metric multidimensional scaling. In addition, for each taxa significant difference between sample groups will be assessed by comparing the relative number of reads.

SECONDARY OUTCOMES:
fMRI BOLD activity memory performance | 14 days
positive and negative affect | 14 days
  PANAS (Positive and Negative Affect Schedule); scores can range from 10 - 50, with higher (lower) scores representing higher (lower) levels of positive (negative) affect
mood | 14 days
  POMS (Profile of Mood States); four scales (Depression/Anxiety, Fatigue, Vigor, Anger), 35 items, 7 point scale, instruction "How you have been feeling during the past 24 hours?"
emotional health | 14 days
  BDI-II (Beck Depression Inventory); score minimum 0 to maximum 21
well-being | 14 days
  WHO-5 (World Health Organization Well-Being Index); measures life quality and life contentment; score minimum 0 to maximum 5 with higher score representing higher life quality and life contentment
satiety | 14 days
  self-reported hunger scale; visual analogue scale; score minimum 0 to maximum 8
serum lipid metabolism markers | 14 days
  total cholesterol, triglycerides, high density lipoprotein, low density lipoprotein
serum glucose metabolism markers | 14 days
  glucose, insulin
serum glucose metabolism markers | 14 days
  long-term glucose marker HbA1C
serum inflammatory markers | 14 days
  high sensitivity C-reactive protein, interleukin-6
hunger hormones | 14 days
  leptin, ghrelin, Glucagon-like peptide-1 (GLP-1), peptide YY
serum microbial metabolic markers | 14 days
  short-chain fatty acids (SCFA), trimethylamine N-oxide (TMAO), bile acids
personality traits | 14 days
  BFMM (BIG FIVE Mine Marker); measures the Big Five personality traits as states; 5 subscales (neuroticism, extraversion, openness, agreeableness, conscientiousness); higher scores means being more extreme for a certain state
gastrointestinal health | 14 days
  GQLI-10 (Gastrointestinal Quality of Life Index); 10 items to measure quality of life regarding gastrointestinal symptoms; the higher the score the stronger the symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Max Planck Institute for Human Cognitive and Brain Sciences, Leipzig, Saxony, Germany

REFERENCES:
- [Derived] Medawar E, Beyer F, Thieleking R, Haange SB, Rolle-Kampczyk U, Reinicke M, Chakaroun R, von Bergen M, Stumvoll M, Villringer A, Witte AV. Prebiotic diet changes neural correlates of food decision-making in overweight adults: a randomised controlled within-subject cross-over trial. Gut. 2024 Jan 5;73(2):298-310. doi: 10.1136/gutjnl-2023-330365. PMID 37793780
- [Derived] Medawar E, Haange SB, Rolle-Kampczyk U, Engelmann B, Dietrich A, Thieleking R, Wiegank C, Fries C, Horstmann A, Villringer A, von Bergen M, Fenske W, Veronica Witte A. Gut microbiota link dietary fiber intake and short-chain fatty acid metabolism with eating behavior. Transl Psychiatry. 2021 Oct 1;11(1):500. doi: 10.1038/s41398-021-01620-3. PMID 34599144